CLINICAL TRIAL: NCT01826838
Title: A Phase I Study of Dasatinib, Androgen Deprivation Therapy and Radiation For Intermediate and High Risk Prostate Cancer
Brief Title: Study of Dasatinib, Androgen Deprivation Therapy and Radiation
Acronym: BrUOGPR255
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 255
Record Dates: First submitted 2012-07-24; First posted 2013-04-09 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Three dasatinib dose levels will be evaluated, 50 mg/day, 70 mg/day and 100 mg/day. Dasatinib will begin with day #1 of radiation and will be discontinued once radiation is completed.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — 1.1 Primary Objective 1.1.1 To evaluate the maximum tolerated dose and dose limiting toxicities of dasatinib, up to a dose of 100mg/day, with concurrent standard radiation and hormone therapy for patients with intermediate and high risk prostate cancer.
  1.2 Secondary Objective: 1.2.1 To determine the time to progression and overall survival for patients who are diagnosed with Intermediate and High Risk Prostate Cancer and were treated with dasatinib.

SUMMARY:
Radiation and androgen deprivation is a common modality for patients with localized prostate cancer. Unfortunately for patients with intermediate to high risk prostate cancer incomplete tumor eradication and subsequent relapse occurs in 50-75% of patients. The Src pathway appears to be integral to the pathobiology of prostate cancer and may be fundamental to radioresistance.

DETAILED DESCRIPTION:
Radiation and androgen deprivation is a common modality for patients with localized prostate cancer. Unfortunately for patients with intermediate to high risk prostate cancer incomplete tumor eradication and subsequent relapse occurs in 50-75% of patients. The Src pathway appears to be integral to the pathobiology of prostate cancer and may be fundamental to radioresistance.

The primary objective of this trial will be to establish the safety of dasatinib with androgen deprivation and radiation for prostate cancer. Three dasatinib dose levels will be evaluated, 50 mg/day, 70 mg/day and 100 mg/day. Dasatinib will begin with day #1 of radiation and will be discontinued once radiation is completed. The study treatment period, therefore, will be when patients receive concurrent dasatinib, hormone therapy and radiation to 30 days after the last radiation/dasatinib treatment. However, it will be highly recommended that, prior to entering the study, patients receive 2 months of androgen deprivation with a LHRH agonist. Furthermore, it will be highly recommended that, after completion of dasatinib /hormone therapy/radiation, patients with intermediate risk disease receive approximately 2 additional months of hormone therapy (to complete 6 months of hormone therapy) and patients with high risk disease receive 20 additional months of ADT to complete 2 years of hormone therapy. If casodex was given at onset of diagnosis, patient must be off drug for 6 weeks prior to beginning radiation therapy

ELIGIBILITY:
PATIENT ELIGIBILITY

-Conditions for Patient Eligibility

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Histologically or pathologically confirmed adenocarcinoma of the prostate to be treated with radiation therapy and hormone therapy.
* Intermediate, high or very high risk disease

  * Intermediate-risk disease (clinical T2b or T2c stage or PSA 10 to 20 ng/mL or Gleason score 7)
  * High-risk disease (Gleason score 8 to 10, serum PSA > 20 ng/mL or T3a disease)
  * Very high-risk disease (T3b or T4)
* No prior pelvic or prostate radiation or chemotherapy for prostate cancer.
* Clinically negative lymph nodes as established by imaging (pelvic CT or pelvic MR), nodal sampling or dissection within 8 weeks prior to registration. Patients with lymph nodes equivocal or questionable by imaging are eligible if the nodes are < 1.5 cm.
* Bone scan within 12 weeks prior to registration. Equivocal bone scan findings are allowed if plain films are negative for metastasis.
* ECOG performance status 0-1
* Age > 18
* Required entry laboratory parameters within 14 days of study entry: Granulocytes ≥ 1500/µl; platelet count ≥ 100,000/µl; Hgb > 8.0 g/dl; Creatinine < 1.5 x the institutional ULN, mg/dl; Bilirubin ≤ 2x institutional upper limit of normal; AST ≤ 2.5 x upper limit of normal, Serum Na+, K+, Mg2+, Phosphate and Calcium within institutional normal range; PT and PTT < 1.5 ULN
* Life expectancy of at least 1 year
* No concurrent anticancer therapy.
* Peripheral neuropathy must be ≤ Grade 2
* A male subject of fathering potential must use an adequate method of contraception throughout the study [and for at least 4 weeks after the last dose of study drug].
* Ability to take oral medication (dasatinib must be swallowed whole)
* Signed study-specific consent form prior to study entry

Conditions for Patient Ineligibility

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Evidence of distant metastases (M1).
* Prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy for any reason
* PSA > 150
* Pathologically positive lymph nodes or nodes > 1.5 cm on imaging
* Major medical or psychiatric illness which, in the investigator's opinion, would prevent completion of treatment and would interfere with follow-up.
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable.
* Prior radiotherapy, including brachytherapy, to the region of the study cancer that would result in overlap of radiation therapy fields
* Medical History and Concurrent Diseases
* No malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years.
* Concurrent medical condition which may increase the risk of toxicity, including:
* Pleural or pericardial effusion of any grade
* Cardiac Symptoms; any of the following should be considered for exclusion:
* History of significant bleeding disorder unrelated to cancer, including:
* No history of pulmonary hypertension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of dasatinib with concurrent standard radiation and hormone therapy | 3 months
  Maximum tolerated dose of dasatinib with concurrent standard radiation and hormone

SECONDARY OUTCOMES:
Time to progression for patients | 12 weeks
  Time to progression for patients

CONTACTS AND LOCATIONS:
Overall Officials: anthony mega, Principal Investigator — Brown University